CLINICAL TRIAL: NCT03730883
Title: The Effect of Early Versus Standard Central Line Removal on Growth of Very Low Birth Weight Premature Infants: A Non-inferiority, Randomized Controlled Trial
Brief Title: The Effect of Early Versus Standard Central Line Removal on Growth of Very Low Birth Weight Premature Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Princess Anna Mazowiecka Hospital, Warsaw, Poland (Other)
Collaborators: Nutricia Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CLAG'18
Record Dates: First submitted 2018-11-01; First posted 2018-11-05 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-01

CONDITIONS: Growth Failure; CLABSI - Central Line Associated Bloodstream Infection
MeSH Terms: conditions — Failure to Thrive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Central line removal at 100ml/kg/day. (Experimental): In this group central line will be removed at the time the infant reaches 100 ml/kg/day of enteral intake. Central lines will be removed after 3 well tolerated consecutive feedings (assessed by the physician) with no contraindications for central line removal present.
  Assessment of feedings tolerance will be at discretion of the physician taking care for the infant. After central line removal, infants in this group may continue to receive parenteral nutrition via peripheral venous access, depending on the decision of the physician taking care for the infant.
  Parenteral nutrition will be prescribed according to the local protocol. Enteral nutrition will be initiated during the first days of life and advanced gradually at the discretion of the neonatologist.
  Interventions: Procedure: Central line removal at 100ml/kg/day.
- Central line removal at 140 ml/kg/day. (Active Comparator): In this group central line will be removed at the time the infant reaches 140 ml/kg/day of enteral intake (full enteral intake). In this group central line will be removed at the time the infant reaches 100 ml/kg/day of enteral intake. Central lines will be removed after 3 well tolerated consecutive feedings (assessed by the physician) with no contraindications for central line removal present.
  Assessment of feedings tolerance will be at discretion of the physician taking care for the infant.
  Parenteral nutrition will be prescribed according to the local protocol. Enteral nutrition will be initiated during the first days of life and advanced gradually at the discretion of the neonatologist.
  Interventions: Procedure: Central line removal at 140ml/kg/day.

INTERVENTIONS:
Procedure: Central line removal at 100ml/kg/day. — In this group central line will be removed at the time the infant reaches 100 ml/kg/day of enteral intake if well tolerated.
  Arms: Central line removal at 100ml/kg/day.
Procedure: Central line removal at 140ml/kg/day. — In this group central line will be removed at the time the infant reaches 140 ml/kg/day of enteral intake if well tolerated.
  Arms: Central line removal at 140 ml/kg/day.

SUMMARY:
This study compares two different regimens of a central line removal in respect to weight at 36 weeks postmenstrual age in very low birth weight (VLBW) preterm infants. Half of participants will have a central line removed at ≥100 ml/kg/d, while the other half will have a central line removed at ≥ 140 ml/kg/day.

DETAILED DESCRIPTION:
Eligible infants will be randomized in equal proportions between two groups. In the first group (group A - early central line removal) central line will be removed at the time the infant reaches 100 ml/kg/d of enteral intake. In the second group (group B - standard central line removal) central line will be removed at the time the infant reaches 140 ml/kg/d of enteral intake (full enteral intake). Central lines will be removed after 3 well tolerated consecutive feedings (assessed by the physician) with no contraindications for central line removal present:

* necessity of administration of drugs that must be given via central venous access,
* necessity of administration of drugs that must be given intravenously along with difficulties to secure peripheral venous access,
* necessity of prolonged (> 7 days) administration of drugs that must be given intravenously,
* necessity to continue parenteral nutrition along with difficulties to secure peripheral venous access.

Assessment of feedings tolerance will be at discretion of the physician taking care for the infant. After central line removal, infants in group A will continue to receive parenteral nutrition via peripheral venous access at the discretion of the physician taking care for the infant. The solution used to continue parenteral nutrition via peripheral venous access will contain at maximum 2,5% amino acids, 10% glucose and no calcium or phosphate preparations to ensure fluid's osmolality will not exceed 900 mOsm/l and the solution will be well tolerated when administered via peripheral vein.

Parenteral nutrition will be prescribed according to the local protocol. Enteral nutrition will be initiated during the first days of life and advanced gradually at the discretion of the neonatologist.

ELIGIBILITY:
Inclusion Criteria:

1. Birth weight ≤ 1500 g (very low birth weight).
2. Birth weight ≥ 3rd percentile at a given gestational age.
3. Central line inserted (PICC or UVC).
4. Oral intake not exceeding 100 ml/kg/d at randomization.
5. Lack of congenital illness or malformation that may affect growth.
6. Signed parental consent.

Exclusion Criteria:

1. Birth weight > 1500 g.
2. Birth weight < 3rd percentile at a given gestational age.
3. The absence of a central line.
4. Oral intake ≥100 ml/kg/d at randomization.
5. Congenital illness or malformation that may affect growth.
6. Lack of informed consent.
7. Participation in other intervention (investigational) trials, that may affect the primary outcome.

Max Age: 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 214 (Actual)
Dates: Start 2019-01-26 (Actual); Primary Completion 2022-04-10 (Actual); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Weight at 36 weeks PMA. | 36 weeks PMA.
  Difference between the two intervention arms in weight at 36 weeks PMA. Noninferiority would be declared if a mean difference in weight at 36 weeks PMA will be no more than 210 g.

SECONDARY OUTCOMES:
Head circumference at 36 weeks PMA. | 36 weeks PMA.
  Difference between the two intervention arms in head circumference at 36 weeks PMA.
Length at 36 weeks PMA. | 36 weeks PMA.
  Difference between the two intervention arms in length at 36 weeks PMA.
The rate of CLABSI. | From enrollment up to 2 days after central line removal; day of central line removal is considered Day 1.
  The rate of CLA-BSI in both groups.
Time to regain birth weight. | Up to 4 weeks.
  If the infants remain above their birth weight for 3 consecutive days, the first day of the 3 weights will be used as the date of regaining birth weight.
Number of peripheral intravenous accesses inserted until discontinuation of parenteral nutrition. | Up to 7 days post-intervention.
  Safety of early central line removal will be assessed in respect to number of peripheral intravenous accesses inserted until discontinuation of parenteral nutrition.
Central line insertion due to feeding intolerance. | Up tp 7 days post-intervention.
  Need for central line insertion within 7 days following intervention because of feeding intolerance.
Weight at 18 to 22 months corrected age (CA). | At 18 to 22 months corrected age (CA).
  Weight at the age of 18 to 22 months corrected age (CA) will be assessed for noninferiority.
Length at 18 to 22 months corrected age (CA). | At 18 to 22 months corrected age (CA)
  Length at the age of 18 to 22 months corrected age (CA) will be assessed for noninferiority.
Head circumference at 18 to 22 months corrected age (CA). | At 18 to 22 months corrected age (CA).
  Head circumference at the age of 18 to 22 months corrected age (CA) will be assessed for noninferiority.
Length of hospital stay. | Through study completion, an average of 2 years.
  The data on the length of hospital stay expressed in days will be recorded.

OTHER OUTCOMES:
Growth velocity. | From birth to 36 weeks' PMA.
  Growth velocity will be calculated using exponential method. This outcome will be assessed for noniferiority.
Z-score for weight at birth. | Through study completion, an average of 4 months.
  Z-scores for weight at birth will be compared between the two study groups. We will use Fenton 2013 dataset to determine Z-scores.
Z-score for head circumference at birth. | Through study completion, an average of 4 months.
  Z-scores for head circumference at birth will be compared between the two study groups. We will use Fenton 2013 dataset to determine Z-scores.
Z-score for weight at 36 weeks' PMA. | Through study completion, an average of 4 months.
  Z-scores for weight at 36 weeks' PMA will be compared between the two study groups. We will use Fenton 2013 dataset to determine Z-scores.
Z-score for head circumference at 36 weeks' PMA. | Through study completion, an average of 4 months.
  Z-scores for head circumference at 36 weeks' PMA will be compared between the two study groups. We will use Fenton 2013 dataset to determine Z-scores.
Change in Z-score for weight from birth to 36 weeks' PMA. | Through study completion, an average of 4 months.
  Changes in Z-scores for weight from birth to 36 weeks' PMA will be compared between the two study groups. We will use Fenton 2013 dataset to determine Z-scores.
Change in Z-score for head circumference from birth to 36 weeks' PMA. | Through study completion, an average of 4 months.
  Changes in Z-scores for head circumference from birth to 36 weeks' PMA will be compared between the two study groups. We will use Fenton 2013 dataset to determine Z-scores.

CONTACTS AND LOCATIONS:
Overall Officials: Justyna Romanska, MD, Principal Investigator — Department of Neonatology and Neonatal Intensive Care Warsaw Medical University
Locations (4):
- Poland (4):
  - Department of Neonatology and Neonatal Intensive Care Warsaw Medical University, Warsaw
  - Department of Reproductive Health, Centre of Postgraduate Medical Education, Warsaw
  - Division of Neonatology and Neonatal Intensive Care, 1st Department of Obstetrics and Gynaecology, The Medical University of Warsaw, Warsaw
  - Department of Neonatology, Wroclaw Medical University, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be available, after deidentiﬁcation. The study protocol will also be available. These documents will be accessible to anyone who provides a methodologically sound proposal immediately following publication with no end date.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who provides a methodologically sound proposal.

REFERENCES:
- [Background] Poindexter B. Approaches to growth faltering. World Rev Nutr Diet. 2014;110:228-38. doi: 10.1159/000358471. Epub 2014 Apr 11. PMID 24751633
- [Background] Sengupta A, Lehmann C, Diener-West M, Perl TM, Milstone AM. Catheter duration and risk of CLA-BSI in neonates with PICCs. Pediatrics. 2010 Apr;125(4):648-53. doi: 10.1542/peds.2009-2559. Epub 2010 Mar 15. PMID 20231192
- [Background] Stephens BE, Walden RV, Gargus RA, Tucker R, McKinley L, Mance M, Nye J, Vohr BR. First-week protein and energy intakes are associated with 18-month developmental outcomes in extremely low birth weight infants. Pediatrics. 2009 May;123(5):1337-43. doi: 10.1542/peds.2008-0211. PMID 19403500
- [Background] Dusick AM, Poindexter BB, Ehrenkranz RA, Lemons JA. Growth failure in the preterm infant: can we catch up? Semin Perinatol. 2003 Aug;27(4):302-10. doi: 10.1016/s0146-0005(03)00044-2. PMID 14510321
- [Background] Ehrenkranz RA, Dusick AM, Vohr BR, Wright LL, Wrage LA, Poole WK. Growth in the neonatal intensive care unit influences neurodevelopmental and growth outcomes of extremely low birth weight infants. Pediatrics. 2006 Apr;117(4):1253-61. doi: 10.1542/peds.2005-1368. PMID 16585322
- [Background] Ibrahim HM, Jeroudi MA, Baier RJ, Dhanireddy R, Krouskop RW. Aggressive early total parental nutrition in low-birth-weight infants. J Perinatol. 2004 Aug;24(8):482-6. doi: 10.1038/sj.jp.7211114. PMID 15167885
- [Background] Stoll BJ, Hansen NI, Adams-Chapman I, Fanaroff AA, Hintz SR, Vohr B, Higgins RD; National Institute of Child Health and Human Development Neonatal Research Network. Neurodevelopmental and growth impairment among extremely low-birth-weight infants with neonatal infection. JAMA. 2004 Nov 17;292(19):2357-65. doi: 10.1001/jama.292.19.2357. PMID 15547163
- [Background] Alshaikh B, Yee W, Lodha A, Henderson E, Yusuf K, Sauve R. Coagulase-negative staphylococcus sepsis in preterm infants and long-term neurodevelopmental outcome. J Perinatol. 2014 Feb;34(2):125-9. doi: 10.1038/jp.2013.155. Epub 2013 Dec 19. PMID 24355942
- [Background] Donovan EF, Sparling K, Lake MR, Narendran V, Schibler K, Haberman B, Rose B, Meinzen-Derr J; Ohio Perinatal Quality Collaborative. The investment case for preventing NICU-associated infections. Am J Perinatol. 2013 Mar;30(3):179-84. doi: 10.1055/s-0032-1322516. Epub 2012 Jul 26. PMID 22836823
- [Background] O'Grady NP, Alexander M, Burns LA, Dellinger EP, Garland J, Heard SO, Lipsett PA, Masur H, Mermel LA, Pearson ML, Raad II, Randolph AG, Rupp ME, Saint S; Healthcare Infection Control Practices Advisory Committee. Guidelines for the prevention of intravascular catheter-related infections. Am J Infect Control. 2011 May;39(4 Suppl 1):S1-34. doi: 10.1016/j.ajic.2011.01.003. No abstract available. PMID 21511081
- [Background] Milstone AM, Reich NG, Advani S, Yuan G, Bryant K, Coffin SE, Huskins WC, Livingston R, Saiman L, Smith PB, Song X. Catheter dwell time and CLABSIs in neonates with PICCs: a multicenter cohort study. Pediatrics. 2013 Dec;132(6):e1609-15. doi: 10.1542/peds.2013-1645. Epub 2013 Nov 11. PMID 24218474
- [Background] Fisher D, Cochran KM, Provost LP, Patterson J, Bristol T, Metzguer K, Smith B, Testoni D, McCaffrey MJ. Reducing central line-associated bloodstream infections in North Carolina NICUs. Pediatrics. 2013 Dec;132(6):e1664-71. doi: 10.1542/peds.2013-2000. Epub 2013 Nov 18. PMID 24249819
- [Background] Drenckpohl D, McConnell C, Gaffney S, Niehaus M, Macwan KS. Randomized trial of very low birth weight infants receiving higher rates of infusion of intravenous fat emulsions during the first week of life. Pediatrics. 2008 Oct;122(4):743-51. doi: 10.1542/peds.2007-2282. PMID 18829797
- [Derived] Romanska J, Margas W, Bokiniec R, Krajewski P, Seliga-Siwecka J. Effect of early versus standard central line removal on growth of very low birthweight premature infants: a protocol for a non-inferiority randomised controlled trial. BMJ Open. 2019 Sep 17;9(9):e030167. doi: 10.1136/bmjopen-2019-030167. PMID 31530607
- See also: IHI - How-to Guide: Prevent Central Line-Associated Bloodstream Infections. Cambridge, MA: Institute for Healthcare Improvement; 2012 — http://www.ihi.org/
- See also: International Fetal and Newborn Growth Standards for the 21st Century. Anthropometry Handbook. University of Oxford; 2012 — https://www.medscinet.net/Intergrowth/patientinfodocs/Anthropometry%20Handbook%20April%202012.pdf
- See also: Nutritional Support of the Very Low Birth Weight Infant. Toolkit Rev.2018. — https://www.cpqcc.org/
- See also: Centers for Disease Control and Prevention. Central Line-Associated Bloodstream Infection (CLABSI) Event. — https://www.cdc.gov/nhsn/PDFs/pscManual/4PSC_CLABScurrent.pdf